CLINICAL TRIAL: NCT02374138
Title: Improving Asthma Outcomes Through Stress Management
Brief Title: Breathe With Ease: A Unique Approach to Managing Stress (BEAMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen J. Teach, MD, MPH (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Stephen J. Teach, MD, MPH, Chair, Pediatrics, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5819
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Asthma
Keywords: psychosocial stress
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): IMPACT DC Asthma Clinic intervention of guideline-based clinical care, education, and short-term care coordination
  Interventions: Other: Usual Care
- Intervention (Experimental): Parental stress management in addition to IMPACT DC intervention of guideline-based clinical care, education, and short-term care coordination.
  Interventions: Behavioral: Parental stress management

INTERVENTIONS:
Behavioral: Parental stress management — The intervention for this study is a multi-dimensional stress management program designed to be responsive to parent and other stakeholder preferences. The intervention will have two separate yet coordinated components: one-on-one stress management sessions and peer group sessions led by "community wellness coaches."
  Arms: Intervention
Other: Usual Care — IMPACT DC Asthma Clinic intervention of guideline-based clinical care, education, and short-term care coordination
  Arms: Usual Care

SUMMARY:
Uncontrolled asthma in at-risk youth responds well to guideline-based therapy when patients remain adherent to their management plans. Adherence to inhaled corticosteroids (ICS), when indicated for persistent or uncontrolled asthma, is a critical component of most asthma management plans, and other self-management practices such as trigger avoidance are similarly related to improved asthma outcomes. Adherence to self-management practices is mediated by multiple factors, including psychosocial stress of parents and their children.

A targeted, culturally appropriate intervention to manage psychosocial stress among the parents of young, African American, and socioeconomically disadvantaged urban children with asthma who are receiving guideline-based care may improve asthma self-management, and therefore asthma outcomes.

Our overall aim is to implement and evaluate a highly collaborative, multi-dimensional, culturally appropriate and community-based asthma intervention to augment existing guideline-based best practice. The intervention will target the parents of at-risk, urban, African American youth, and will employ individualized psychosocial stress management and peer support.

DETAILED DESCRIPTION:
Uncontrolled asthma in at-risk youth responds well to guideline-based therapy when patients remain adherent to their management plans. Adherence to inhaled corticosteroids (ICS), when indicated for persistent or uncontrolled asthma, is a critical component of most asthma management plans, and other self-management practices such as trigger avoidance are similarly related to improved asthma outcomes. Adherence to self-management practices is mediated by multiple factors, including psychosocial stress of parents and their children.

A targeted, culturally appropriate intervention to manage psychosocial stress among the parents of young, African American, and socioeconomically disadvantaged urban children with asthma who are receiving guideline-based care may improve asthma self-management, and therefore asthma outcomes.

Our overall aim is to implement and evaluate a highly collaborative, multi-dimensional, culturally appropriate and community-based asthma intervention to augment existing guideline-based best practice. The intervention will target the parents of at-risk, urban, African American youth, and will employ individualized psychosocial stress management and peer support.

We will conduct a single blind, prospective randomized controlled trial comparing the IMPACT DC Asthma Clinic's existing intervention of guideline-based clinical care, education, and short-term care coordination (usual care) to usual care plus parental stress management in a cohort of up to 200 parent-child dyads of AA youth aged 4-12 years.

ELIGIBILITY:
We plan to enroll parent-child dyads that meet the following criteria:

Inclusion criteria (Parent):

* self-identify as African-American
* both the legal guardian and primary asthma caregiver of an eligible child.

Exclusion criteria (Parent):

* unable or unwilling to sign informed consent document
* exclusionary psychiatric condition, including but not limited to psychosis, based on the screening form at recruitment
* enrolled in another asthma research study.

Inclusion criteria (Child):

* parent-identified as African-American
* age 4-12 years inclusive at recruitment
* physician diagnosis of persistent asthma
* publicly financed insurance

Exclusion criteria (Child):

- chronic medical condition (other than asthma) including but not limited to diabetes, sickle cell disease, heart disease, lung disease or neurological disorder.

In addition, the PI may choose to not include a participant if he does not believe it is in the family's best interest to participate.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Teach, MD, MPH, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Teach SJ, Shelef DQ, Foushee N, Horn IB, Yadav K, Wang Y, Rand CS, Streisand R. Randomized clinical trial of parental psychosocial stress management to improve asthma outcomes. J Asthma. 2021 Jan;58(1):121-132. doi: 10.1080/02770903.2019.1665063. Epub 2019 Sep 23. PMID 31545115

RESULTS

PARTICIPANT FLOW:
Period: Six Month Follow Up
Arm/Group | Usual Care | Intervention
Started | 110 | 107
Completed | 102 (6 Month Follow Up) | 93 (6 Month Follow Up)
Not Completed | 8 | 14
Period: Twelve Month FollowUp
Arm/Group | Usual Care | Intervention
Started (All participants were contacted at 12m, regardless of whether they completed the 6m interview.) | 110 | 107
Completed | 101 | 95
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 110 | 107 | 217
Age, Categorical [Count of Participants; unit: Participants]
  Parent Participants: <=18 years | 0 | 0 | 0
  Parent Participants: Between 18 and 65 years | 108 | 104 | 212
  Parent Participants: >=65 years | 2 | 3 | 5
  Child Participants: <=18 years | 110 | 107 | 217
  Child Participants: Between 18 and 65 years | 0 | 0 | 0
  Child Participants: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Parent Participants | 33.2 (8.9) | 34.3 (10.0) | 33.8 (9.5)
  Child Participants | 6.4 (2.3) | 6.8 (2.3) | 6.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Parent Participants: Female | 100 | 100 | 200
  Parent Participants: Male | 10 | 7 | 17
  Child Participants: Female | 42 | 43 | 85
  Child Participants: Male | 68 | 64 | 132
Region of Enrollment [Number; unit: participants]
  United States | 110 | 107 | 217

OUTCOME MEASURES:

1. Primary Outcome: Symptom-free Days in the Last 14 Days
Description: Symptom-free days are defined as a 24-hour period with no coughing, wheezing, chest tightness, or shortness of breath and no need for rescue medications
Time Frame: Repeated Measures at 6 months (3 month data collected to allow for repeated measures)
Population: Randomized participants with follow up available at each time period.
Measure: Mean (Standard Deviation); unit: days in prior 14d
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
days in prior 14d | 11.4 (3.3) | 11.6 (3.0)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; At 6 Months; Test type: Superiority; p = 0.93, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender

2. Secondary Outcome: Asthma Morbidity - Nighttime Asthma Symptoms
Description: Nights of asthma symptoms in prior 14d
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants with data available at each follow up time point
Measure: Mean (Standard Deviation); unit: days in prior 14d
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
days in prior 14d
  Nighttime asthma symptoms at 6 Month FU: number analyzed (Participants) | 102 | 93
  Nighttime asthma symptoms at 6 Month FU | 1.7 (2.9) | 1.9 (3.2)
  Nighttime asthma symptoms at 12 Month FU: number analyzed (Participants) | 101 | 95
  Nighttime asthma symptoms at 12 Month FU | 2.1 (3.2) | 1.5 (2.3)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; At 6 month follow up; Test type: Superiority; p = 0.87, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; At 12 month follow up; Test type: Superiority; p = 0.25, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender

3. Secondary Outcome: Asthma Severity and Control
Time Frame: Repeated Measures at 3, 6, and 12 months
Population: Data not collected
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Asthma Medication Adherence
Description: Reported use of inhaled corticosteroids and LTRA in past two days
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants with Follow Up Data Available at Each Time Point
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  ICS use at 6 Month Follow Up: number analyzed (Participants) | 102 | 93
  ICS use at 6 Month Follow Up | 68 | 68
  ICS use at 12 Month Follow up: number analyzed (Participants) | 101 | 95
  ICS use at 12 Month Follow up | 55 | 61
  LTRA use at 6 Month Follow Up: number analyzed (Participants) | 102 | 93
  LTRA use at 6 Month Follow Up | 14 | 16
  LTRA use at 12 Month Follow Up: number analyzed (Participants) | 101 | 95
  LTRA use at 12 Month Follow Up | 20 | 18
Statistical Analysis 1: Comparison: Usual Care vs Intervention; ICS Use at 6 Month Follow Up; Test type: Superiority; p = 0.35, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; ICS Use at 12 Month Follow Up; Test type: Superiority; p = 0.34, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender
Statistical Analysis 3: Comparison: Usual Care vs Intervention; LTRA Use at 6 Months; Test type: Superiority; p = 0.35, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender
Statistical Analysis 4: Comparison: Usual Care vs Intervention; LTRA use at 12 Month Follow Up; Test type: Superiority; p = 0.62, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender

5. Secondary Outcome: Health Care Utilization - Emergency Department Visits for Asthma
Description: Health care utilization - emergency department visits for asthma over six month and twelve month follow up periods. Reported as those documented in the electronic medical record of Children's National Health System plus parent report of visits elsewhere
Time Frame: 12 months after enrollment
Population: Participants with follow up available at each time point
Measure: Mean (Standard Error); unit: Visits
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Visits
  ED Visits between enrollment and 6m Follow Up: number analyzed (Participants) | 102 | 93
  ED Visits between enrollment and 6m Follow Up | 0.32 (0.68) | 0.32 (0.77)
  ED Visits between 6m and 12m Follow up: number analyzed (Participants) | 101 | 95
  ED Visits between 6m and 12m Follow up | 0.33 (0.65) | 0.42 (0.75)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; ED visits over 6 months; Test type: Superiority; p = 0.63, Generalized Linear Model Analysis — Adjusted for child age, gender, and baseline value
Statistical Analysis 2: Comparison: Usual Care vs Intervention; ED Visits between 6 and 12 Month follow up; Test type: Superiority; p = 0.44, Generalized Linear Model Analysis — Adjusted for child age, gender, and baseline value

6. Secondary Outcome: Asthma Exacerbations - Courses of Systemic Steroids
Description: Courses of systemic steroids over 12m follow up period
Time Frame: Assessed at 6m and 12m following enrollment
Population: Participants with data available at each time point
Measure: Mean (Standard Error); unit: Courses of systemic steroids
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Courses of systemic steroids
  Courses of systemic steroids over 6 Months: number analyzed (Participants) | 102 | 93
  Courses of systemic steroids over 6 Months | 0.30 (0.63) | 0.29 (0.68)
  Courses of systemic steroids btwn 6m and 12m FU: number analyzed (Participants) | 101 | 95
  Courses of systemic steroids btwn 6m and 12m FU | 0.26 (0.61) | 0.30 (0.67)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Courses of systemic steroids over 6 months; Test type: Superiority; p = 0.98, Generalized Linear Model Analysis — Adjusted for child age, gender, and baseline value
Statistical Analysis 2: Comparison: Usual Care vs Intervention; Courses of systemic steroids between 6m and 12m FU; Test type: Superiority; p = 0.48, Generalized Linear Model Analysis — Adjusted for child age, gender, and baseline value

7. Secondary Outcome: Parental Stress
Description: Score on Perceived Stress Scale (PSS). The Perceived Stress Scale consists of 10 questions and is a measure of the degree to which situations in one's life are appraised as stressful. Scores range from 0 - 40, with higher scores indicating a higher level of perceived stress.
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Number of participants with follow up available at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale
  PSS Score at 6 Month Follow Up: number analyzed (Participants) | 102 | 93
  PSS Score at 6 Month Follow Up | 10.4 (7.3) | 11.4 (7.1)
  PSS Score at 12 Month Follow up: number analyzed (Participants) | 101 | 95
  PSS Score at 12 Month Follow up | 10.3 (7.2) | 12.6 (7.8)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; At 6 Month Follow Up; Test type: Superiority; p = 0.32, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; At 12 Month Follow Up; Test type: Superiority; p = 0.06, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender

8. Secondary Outcome: Parental Depression
Description: Score on Center for Epidemiologic Studies Depression Scale (CES-D - 10). The CESD-10 scale screens for depressive symptoms. Scores range from 0-30, with higher scores indicating a higher degree of depressive symptoms.
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants available at each follow up time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale
  CES-D 10 score at 6 Month Follow up: number analyzed (Participants) | 102 | 93
  CES-D 10 score at 6 Month Follow up | 6.8 (4.8) | 7.4 (5.2)
  CES-D 10 score at 12 Month Follow up: number analyzed (Participants) | 101 | 95
  CES-D 10 score at 12 Month Follow up | 7.6 (5.7) | 8.0 (5.8)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; At 6 Month follow up; Test type: Superiority; p = 0.32, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; At 12 month follow up; Test type: Superiority; p = 0.44, Generalized Linear Model Analysis — By repeated measures, p-value adjusted for age and gender

9. Secondary Outcome: Child Anxiety
Description: PROMIS Parent Proxy Anxiety. For PROMIS instruments, T-scores rescale the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher T-score represents higher anxiety and/or depression.
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants available at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale
  Score at 6 Month Follow up: number analyzed (Participants) | 102 | 93
  Score at 6 Month Follow up | 42.5 (9.6) | 40.4 (7.8)
  Score at 12 Month Follow Up: number analyzed (Participants) | 101 | 95
  Score at 12 Month Follow Up | 43.1 (10.2) | 41.5 (8.4)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; At 6 Month Follow Up; Test type: Superiority; p = 0.70, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; At 12 Month Follow Up; Test type: Superiority; p = 0.80, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender

10. Secondary Outcome: Child Depression
Description: PROMIS Parent Proxy Depressive Symptoms is a parent-report assessment of child depression. For PROMIS instruments, T-scores rescale the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher T-score represents higher anxiety and/or depression.
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants available at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale
  Score at 6 Month Follow Up: number analyzed (Participants) | 102 | 93
  Score at 6 Month Follow Up | 41.1 (7.7) | 40.6 (7.0)
  Score at 12 Month Follow Up: number analyzed (Participants) | 101 | 95
  Score at 12 Month Follow Up | 42.3 (9.1) | 41.2 (7.6)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; 6 Month Follow Up; Test type: Superiority; p = 0.53, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; 12 Month Follow up; Test type: Superiority; p = 0.77, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender

11. Secondary Outcome: Caregiver Quality of Life
Description: Caregiver quality of life score, assessed by modified Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ). The measure had five response options, with scores ranging from 13-65 and higher scores meaning better quality of life. No subscales were analyzed.
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants with follow up available at each time point. Note use of modified scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale
  Score at 6 month Follow Up: number analyzed (Participants) | 102 | 93
  Score at 6 month Follow Up | 57.6 (8.8) | 58.9 (8.1)
  Score at 12 Month Follow Up: number analyzed (Participants) | 101 | 95
  Score at 12 Month Follow Up | 58.1 (8.4) | 57.8 (8.4)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Quality of Life at 6 Month Follow up; Test type: Superiority; p = 0.53, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; Quality of Life at 12 Month Follow up; Test type: Superiority; p = 0.57, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender

12. Secondary Outcome: Number of Participants With AEs and SAEs
Description: Safety data: Number of Participants with AEs and SAEs
Time Frame: 12m follow up period
Population: Participants available at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  6 Month Follow Up: number analyzed (Participants) | 102 | 93
  6 Month Follow Up | 0 | 0
  12 Month Follow up: number analyzed (Participants) | 101 | 95
  12 Month Follow up | 0 | 0
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority; p = 1.0, Fisher Exact

13. Secondary Outcome: Economic Outcomes
Description: Analysis of costs of care in both groups
Time Frame: 12m follow-up period
Population: Data were not collected
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Caregiver Smoking Behavior
Description: parent report of cigarettes smoked per day
Time Frame: Repeated Measures at 6 and 12 months
Population: We are unable to analyze or report the data because it was not systematically collected.
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Coping Strategies
Description: Brief COPE
Time Frame: Repeated measures at 12m FU (6m data used for repeated measures)
Population: While we have collected this data, its analysis will be complex and require significant resources. We lack those resources at this time. We may at some point in the future return to this analysis.
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Score on Brief COPE at 12 Months; Test type: Superiority; p = 0.58, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender

16. Secondary Outcome: Mindfulness
Description: Interpersonal Mindfulness in Parenting
Time Frame: Repeated Measures at 6 and 12 months
Population: We are unable to analyze or report the data because it was not systematically collected.
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Parental Resilience
Description: Parental resilience assessed by score on Revised Life Orientation Test (LOT-R) measure. The LOT-R assesses optimism/resilience, and is comprised of 10 questions. Scores range from 0-40, with a higher score indicating a higher level of optimism.
Time Frame: Repeated Measures at 6 and 12 months
Population: Participants with follow up available at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale
  Score on LOT-R at 6 Month Follow Up: number analyzed (Participants) | 102 | 93
  Score on LOT-R at 6 Month Follow Up | 16.1 (3.3) | 16.5 (4.5)
  Score on LOT-R at 12 month Follow Up: number analyzed (Participants) | 101 | 95
  Score on LOT-R at 12 month Follow Up | 16.7 (3.3) | 16.9 (4.1)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Score on LOT-R at 6 Month Follow Up; Test type: Superiority; p = 0.46, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; Score on LOT-R at 12 Month Follow Up; Test type: Superiority; p = 0.62, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender

18. Secondary Outcome: Exacerbations - Hospital Admissions
Description: Number of participants with hospital admissions due to exacerbations
Time Frame: Assessed at 6m and 12m after enrollment
Population: Participants with data available at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  Pts hospitalized btwn enrollment and 6m FU: number analyzed (Participants) | 102 | 93
  Pts hospitalized btwn enrollment and 6m FU | 5 | 4
  Pts hospitalized btwn 6m and 12m FU: number analyzed (Participants) | 101 | 95
  Pts hospitalized btwn 6m and 12m FU | 7 | 9

19. Secondary Outcome: Symptom-free Days in the Last 14 Days
Description: as for outcome 1
Time Frame: Repeated Measures at 12 months (with data also assessed at 3m and 6m)
Population: Participants with data available at 12m follow up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 101 | 95
days | 10.9 (3.7) | 11.8 (2.9)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority — By repeated measures, p-value adjusted for age and gender; p = 0.35, Generalized Linear Model Analysis

20. Secondary Outcome: Asthma Morbidity - Daytime Asthma Symptoms, Days of Activity Limitations, and Days of Quick Relief Medicine Use
Description: Days of asthma symptoms, activity limitation, and quick relief medicine use in prior 14d
Time Frame: Repeated measures at 6 and 12 months (3m data collected for repeated measures)
Population: Participants with data available at each follow up time point
Measure: Mean (Standard Deviation); unit: days in prior 14d
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
days in prior 14d
  Daytime asthma symptoms at 6m FU: number analyzed (Participants) | 102 | 93
  Daytime asthma symptoms at 6m FU | 1.64 (2.48) | 1.83 (2.66)
  Daytime asthma symptoms at 12m FU: number analyzed (Participants) | 101 | 95
  Daytime asthma symptoms at 12m FU | 2.31 (3.24) | 1.57 (2.39)
  Days of activity limitation at 6m: number analyzed (Participants) | 102 | 93
  Days of activity limitation at 6m | 1.42 (2.53) | 1.04 (1.74)
  Days of activity limitation at 12m: number analyzed (Participants) | 101 | 95
  Days of activity limitation at 12m | 1.66 (2.99) | 1.12 (2.31)
  Days of quick relief medicine use at 6m: number analyzed (Participants) | 102 | 93
  Days of quick relief medicine use at 6m | 2.75 (3.59) | 2.96 (4.26)
  Days of quick relief medicine use at 12m: number analyzed (Participants) | 101 | 95
  Days of quick relief medicine use at 12m | 3.40 (4.16) | 2.85 (3.99)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority — Daytime asthma symptoms in prior 14d at 6-month follow up; p = 0.54, Generalized Linear Model Analysis; By repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; Test type: Superiority — Daytime Asthma Symptoms at 12 month follow up; p = 0.11, Generalized Linear Model Analysis; By repeated measures, p-value adjusted for age and gender
Statistical Analysis 3: Comparison: Usual Care vs Intervention; Test type: Superiority — Days of Activity Limitations at 6 month follow up; p = 0.82, Generalized Linear Model Analysis; By repeated measures, p-value adjusted for age and gender
Statistical Analysis 4: Comparison: Usual Care vs Intervention; Test type: Superiority — Days of Activity Limitations at 12 month follow up; p = 0.84, Generalized Linear Model Analysis; By repeated measures, p-value adjusted for age and gender
Statistical Analysis 5: Comparison: Usual Care vs Intervention; Test type: Superiority — Days of Quick Relief Medicine Use at 6 month follow up; p = 0.70, Generalized Linear Model Analysis; By repeated measures, p-value adjusted for age and gender
Statistical Analysis 6: Comparison: Usual Care vs Intervention; Test type: Superiority — Days of Quick Relief Medicine Use at 12 month follow up; p = 0.58, Generalized Linear Model Analysis; By repeated measures, p-value adjusted for age and gender

21. Other Pre Specified Outcome: Sociodemographics
Description: Age, gender, race, ethnicity, insurance type, parental education, household income, family medical history
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  Parent Race : African American | 110 | 107
  Child Race : African American | 110 | 107
  Parent Ethnicity: Non-Hispanic | 110 | 106
  Child Ethnicity: Non-Hispanic | 110 | 106
  Public Insurance | 110 | 107
  Parent Education: Grade 1-11 | 9 | 19
  Parent Education: GED or 12th grade | 44 | 41
  Parent Education: Some college/associates degree | 39 | 33
  Parent Education: College Graduate | 18 | 14
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Parent education; Test type: Other — Univariate test; p = 0.20, Chi-squared

22. Other Pre Specified Outcome: Number of Participants With Positive Smoke Exposure
Description: Participants with environmental smoke exposure. Responses were regrouped as negative (none) or positive (daily, often, or rarely) based on two questions: "How often did anyone smoke inside the home where child usually lives?" or "How often did anyone smoke in the room where child usually sleeps?" A positive response on either or both questions was considered positive exposure.
Time Frame: Repeated Measures at 6 and 12 months (3m data collected for repeated measures)
Population: Number of participants with follow up data available at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  6 Month Follow Up: number analyzed (Participants) | 98 | 89
  6 Month Follow Up | 13 | 10
  12 Month Follow up: number analyzed (Participants) | 101 | 95
  12 Month Follow up | 13 | 9
Statistical Analysis 1: Comparison: Usual Care vs Intervention; ETS exposure at 6 Month Follow Up; Test type: Superiority; p = 0.91, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; ETS Exposure at 12 Month Follow up; Test type: Superiority; p = 0.98, Generalized Linear Model Analysis — Repeated measures, p-value adjusted for age and gender

23. Other Pre Specified Outcome: Parental Health Literacy
Description: Single Item Literacy Screener (SILS)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  Never needs assistance | 98 | 95
  Needs any assistance | 12 | 12
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other — Univariate test; p = 0.94, Chi-squared

24. Other Pre Specified Outcome: Use of Existing Ancillary Services
Time Frame: Assessed at 6m and 12m following enrollment
Population: Participants with data available at each follow up point
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
Participants
  Parent use of mental health resources at 6 Months: number analyzed (Participants) | 101 | 89
  Parent use of mental health resources at 6 Months | 19 | 30
  Parent use of mental health resources at 12 Months: number analyzed (Participants) | 101 | 95
  Parent use of mental health resources at 12 Months | 28 | 28
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Parent use of mental health resources at 6 Months; Test type: Superiority; p = 0.02, Generalized Linear Model Analysis — p-value adjusted for age and gender
Statistical Analysis 2: Comparison: Usual Care vs Intervention; Parent use of mental health resources at 12 Months; Test type: Superiority; p = 0.85, Generalized Linear Model Analysis — p-value adjusted for age and gender

25. Other Pre Specified Outcome: Parental Resilience
Description: as for outcome 17
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 110 | 107
units on a scale | 16.1 (3.3) | 16.2 (3.5)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other — Univariate test; p = 0.90, Wilcoxon (Mann-Whitney)

26. Other Pre Specified Outcome: Intervention Component Uptake
Description: Completion of intervention sessions
Time Frame: 6 month intervention period
Population: Intervention group only
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 107
Participants
  Completed 0 Intervention Sessions | 8
  Completed 1 Intervention Session | 15
  Completed 2 Intervention Sessions | 4
  Completed 3 Intervention Sessions | 5
  Completed 4 Intervention Sessions | 75

27. Other Pre Specified Outcome: Intervention Satisfaction
Description: Brief survey of satisfaction with intervention components.
Time Frame: 6 month intervention period
Population: Participants with data available at 6 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 91
Participants
  "Very Much" satisfied with individual sessions | 82
  "Very Much" satisfied with delivery of sessions | 86

28. Other Pre Specified Outcome: Intervention Fidelity
Description: Checklist of staff's fidelity to individual components of intervention protocol
Time Frame: 6 month intervention period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For duration of trial (12 months following enrollment of each participant)
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/107
Other Adverse Events (participants affected / at risk) | 0/110 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-11-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02374138/SAP_000.pdf
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02374138/Prot_001.pdf